CLINICAL TRIAL: NCT02272543
Title: Acceptability and Efficacy of 'Fish Surimi Peptide' in Under Five Children Suffering From Moderate Acute Malnutrition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Suzuhiro Kamaboko Co., Ltd.,Japan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-14047
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2016-06

CONDITIONS: Moderate Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish surimi peptide powder (Active Comparator): Fish surimi peptide powder
  Interventions: Dietary Supplement: Fish surimi peptide
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Fish surimi peptide

INTERVENTIONS:
Dietary Supplement: Fish surimi peptide

SUMMARY:
Protein-energy malnutrition (PEM) including moderate acute malnutrition (MAM: weight-for-height z-score <-2 to -3, or mid upper arm circumference (MUAC) 115 to < 125 mm) is a major cause of morbidity and mortality in under-5 children of developing/low-income countries. Approximately 14.6% of all under-5 mortality worldwide is attributed to MAM. Prevalence of MAM among under-5 children in Bangladesh is ~12% (~1.7 million). Providing a diet containing adequate nutrients is the mainstay of treatment of children with MAM. Dietary protein is mostly derived from vegetable sources for the middle and low income population among whom the prevalence of MAM and other forms of PEM is high. It is now possible to process fish into fish peptides with longer shelf-life without refrigerator, known as 'fish Surimi' and consumed by different categories of people who need more well-balanced protein; this could be an attractive alternative to supply fish protein in the diet of children in low-income countries like Bangladesh.

Fish Surimi peptide is broken down from white fish meat using plant-derived enzyme and the ingredient is just fish meat consisted of 20 different kinds of amino acids including nine essential amino acids. In human studies it is found to help lowering blood lipids, glucose, IgE, hypertension, and increasing serum albumin and total protein, and bone density.

The present study is designed to assess acceptability and efficacy of 'fish Surimi' in 2-5 years old children suffering from MAM. A pilot study with two phases: to assess the i) acceptability with a small convenience sample (N=30) (phase 1); and ii) efficacy (rate of weight gain) of this fish peptide in a small convenience sample (N=70: 35 intervention 35 control) (phase 2) is proposed.

Acceptability trial (first phase): The investigators will conduct this study in the study ward of Dhaka Hospital of icddr,b. For each child the study will be for two days: i.e. direct observation of food intake of two lunches and two suppers. In a randomly manner and cross over design, an individual child will be offered 5g of fish Surimi during lunch and 5g during supper in one day or the same meal without any fish peptide on the other day in a blinded manner. The investigators will observe the completeness and eagerness of eating and any possible side effect (e.g. allergy, vomiting, diarrhea etc.) over these two days.

Pilot efficacy trial (second phase): The investigators will conduct a pilot trial to assess the efficacy (mainly on child weight gain) of fish Surimi given at home with various foods/meals in 2-5 years old children with MAM will be conducted in Dhaka City of Bangladesh. Children will be enrolled from the Dhaka Hospital of icddr,b after improvement of any acute illness. The intervention group will receive (as take home supplementation) two-week's ration of fish Surimi (@10g/day in two doses i.e. 5g + 5g each in airtight packet), which will be served twice daily mixed with family diet. The control group will not be provided any supplements but the parents will be given dietary advice to provide nutritious food to the child in adequate amounts, and children of both groups will receive micronutrient sprinkle. The child's guardian will be supplied with fish Surimi during initial discharge from icddr,b hospital and requested to come for a fortnightly follow up at the nutrition follow-up unit (NFU) of icddr,b. During each follow-up visit the study research assistant/health worker will do the anthropometry, collect morbidity history since the last visit/follow up and dietary history will also be taken to find out how the child is doing along with the fish Surimi intake. Treatment of any illness will be provided as per standard method by on duty physician of the Dhaka Hospital of icddr,b. The ration for next two weeks will be provided and in such way each child will be followed for ~ 3 months over six NFU-follow-up visits. To reduce the possible drop-out the both-way transportation cost (~ 150 to 250 taka) during each follow-up visit will be reimbursed to the guardians. In the middle of the two scheduled follow-up days the research assistant will call the family by cell phone to monitor the child's feeding and morbidity status. Approximately 5ml blood will be collected from the ante-cubital vein of the children for biochemical test on enrolment and at the end of 3 months and will be analyzed for haemoglobin (Hb), c-reactive protein, zinc, ferritin, albumin, total protein, and IgE. During the blood drawing days each child will be given a toy (take home).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from guardian
* Ages 2 to 5 years
* WHZ<-2 to -3or (MUAC) 115 to < 125 mm without any edema
* Parent/guardian planning to stay in the same area for 3 to 4 months (for smooth follow up purpose)

Exclusion Criteria:

* WHZ ≤ -3 z-scores or presence of bilateral pedal edema
* History of allergy to any fish product
* Anorexia, jaundice or chronic disease or any serious illness warranting hospital referral
* Any congenital anomaly
* Concurrent participation in another clinical trial with intervention to the child

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures: Weight gain after serving the test diet for 12 weeks: changes in body weight during the study period will be measured and 'weight-for-height Z-score 'will be calculated. | 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Azharul Islam Khan, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- icddr,b Dhaka Hospital, Dhaka, Bangladesh